CLINICAL TRIAL: NCT01659294
Title: Impact of Nurse Case Management on Diabetes-related Health Outcomes in a Specialty Care Setting: A Randomized Controlled Trial
Brief Title: Diabetes Outcomes and Nurse Case Manager Study
Acronym: DONCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BCDiabetes.Ca (Network)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Tom Elliott, PI, BCDiabetes.Ca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-Elliott
Record Dates: First submitted 2012-08-02; First posted 2012-08-07 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; outcomes; case management
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nurse case management (Experimental): nurse case management of diabetic variables
  Interventions: Behavioral: Nurse Case Management
- standard diabetologist care (Active Comparator): standard diabetologist care
  Interventions: Behavioral: standard diabetologist care

INTERVENTIONS:
Behavioral: Nurse Case Management
  Arms: nurse case management
Behavioral: standard diabetologist care — routine care by diabetologist & team
  Arms: standard diabetologist care

SUMMARY:
This study will examine whether patients with diabetes who are either 1) newly discharged from hospital or 2) referred to an endocrinologist for management will have better diabetes outcomes when their care is managed primarily by a dedicated case manager (intervention) than by an endocrinologist (standard care) after 6 months of treatment.

DETAILED DESCRIPTION:
The study will be a randomized-control trial recruiting patients with type 2 diabetes in a specialty care setting from two sources:

1. referred by family physicians with inadequate glycemic control likely requiring exogenous insulin therapy
2. referred by medical staff at Vancouver General Hospital or St. Paul's Hospital during in-patient care & about to be discharged (Appendix 1).

Patients who meet the inclusion criteria will be randomly assigned into either the NCM group or SC group.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* A1c > 8.0 or
* BP > 140/90 or
* LDL cholesterol > 2.0 (72 mg/dl)

Exclusion Criteria:

* inability to speak English or to be assisted by somebody fluent in English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
A1c | 6 months
  changes in A1C between NCM vs. SC
diabetes distress (DDS) | 6 months
  changes in diabetes distress between NCM vs. SC. Diabetes Distress (DDS) will be assessed using the 17-item Diabetes Distress Scale (DDS) developed by Polonsky and colleagues. The DDS measures emotional distress and functioning as it relates to living with diabetes. Responses are scored on a 6-point Likert scale (1=no problem to 6=serious problem). A total score is derived by taking the mean of all items. A score of < 2 indicate low/no distress, 2 - 2.9 indicates moderate distress, and score of ≥ 3 indicates high distress.

SECONDARY OUTCOMES:
blood pressure | 6 months
  changes in BP between NCM vs. SC. Blood pressure will be measured using an Omron Digital Blood Pressure Monitor HEM-907. Two upper arm readings are taken with the average of the two recorded.
BMI | 6 months
  changes in BMI between NCM vs. SC. Height and weight will be measured using the Healthometer mechanical eye level upright standard physician scale with attached stadiometer. Body mass index (BMI) are calculated as weight in kilograms divided by height in meters squared.
Self-management behaviours | 6 months
  changes in behaviour habits between NCM vs. SC. Self-management behaviours will be assessed using items from the Summary of Diabetes Self-Care Activities Measure-revised (SDSCA-R).This instrument measures self-care behaviors including diet, exercise, blood sugar testing and foot care. Participants are asked to report the number of days in the past week (range 0-7 days) in which he/she performed specific self-care practices. Greater number of days indicates better self-management.
Medication adherence | 6 months
  changes in medication adherence between NCM vs. SC. Medication adherence will be assessed using the 4-item Moriskyscale that assesses beliefs and behaviors associated with taking medications.Responses are scored on a dichotomous scale: 0=no and 1=yes. A total score is calculated by adding up all items with lower scored indicating better adherence.
Patient motivation | 6 months
  change in patient motivation between NCM vs. SC. motivation will be measured by the 13-item Patient Activation Measure which assesses participants' self-reported knowledge, skills, and confidence an individual has when managing his/her own health.
Diabetes-specific Social Support | 6 months
  change in diabetes-specific social support between NCM vs. SC Diabetes-specific Social Support will be assessed with a 4-item scale developed by Tang et al. that measures amount of support and satisfaction with support from family, friends and the health care team.
Depressive Symptoms Severity | 6 months
  change in depressive symptoms between NCM vs. SC Depressive Symptom Severity will be assessed using the 9-item PRIME-MD Patient Health Questionnaire (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Elliott, MBBS, Principal Investigator — University of British Columbia
Locations (1):
- Bcdiabetes.Ca, Vancouver, British Columbia, Canada

REFERENCES:
- See also: Protocol — https://docs.google.com/open?id=0B9471Ysm3fNqLWdjQy1FVkVDelk
- See also: Consent form — https://docs.google.com/open?id=0B9471Ysm3fNqZDZOMEFncElHRk0